CLINICAL TRIAL: NCT07024667
Title: Clinical and Molecular Study to Evaluate the Effect of the Pixel CO2 Laser (FemiLiftTM) for the Treatment of Vulvo-Vaginal Atrophy (VVA)
Brief Title: Clinical and Molecular Study to Evaluate the Effect of the Pixel CO2 Laser (FemiLiftTM) for the Treatment of Vulvo-Vaginal Atrophy
Acronym: VVA PAP POPQ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0001-21-HYMC
Record Dates: First submitted 2025-05-19; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Vulvar Atrophy; Vaginal Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study intervention group (Experimental): Patients who has vulvo-vaginal atrophy
  Interventions: Device: Pixel CO2 Laser for the Treatment of Vulvo-Vaginal Atrophy (VVA)

INTERVENTIONS:
Device: Pixel CO2 Laser for the Treatment of Vulvo-Vaginal Atrophy (VVA) — Pixel CO2 Laser for the Treatment of Vulvo-Vaginal Atrophy (VVA)

SUMMARY:
Vulvo Vaginal Atrophy (VVA) refers to the changes in the vaginal and vulvar surfaces that occurs during menopause due to the progressive loss of estrogen. The low levels of circulating estrogen produce a wide variety of anatomic, physiologic, and clinical changes in the urogenital area. Clinical symptoms include vaginal dryness, irritation, soreness, dyspareunia, dysuria, and vaginal discharge.

In recent years, microablative fractional CO2 laser has become available for treating vaginal atrophy. It showed a regenerative property with significant histological changes in cellular and connective tissue components. Treatment with the fractional CO2 laser resulted in restoration of the vaginal epithelium with ultrastructural findings, similar to a premenopausal state, that included thickened stratified squamous epithelium with increased collagen support, increased glycogen in epithelial cells, increased fibroblasts, increased vascularity, and presence of sub-epithelial papillae.

DETAILED DESCRIPTION:
Vulvo Vaginal Atrophy (VVA) refers to the changes in the vaginal and vulvar surfaces that occurs during menopause due to the progressive loss of estrogen. The low levels of circulating estrogen produce a wide variety of anatomic, physiologic, and clinical changes in the urogenital area. Clinical symptoms include vaginal dryness, irritation, soreness, dyspareunia, dysuria, and vaginal discharge.

In recent years, microablative fractional CO2 laser has become available for treating vaginal atrophy. It showed a regenerative property with significant histological changes in cellular and connective tissue components. Treatment with the fractional CO2 laser resulted in restoration of the vaginal epithelium with ultrastructural findings, similar to a premenopausal state, that included thickened stratified squamous epithelium with increased collagen support, increased glycogen in epithelial cells, increased fibroblasts, increased vascularity, and presence of sub-epithelial papillae.

The aim of the current study is to evaluate the effect of Pixel CO2 laser, (FemiLiftTM), for the treatment of VVA, on the clinical and molecular levels.

ELIGIBILITY:
Inclusion Criteria:

1. Female 45-75 years of age, at the time of enrolment.
2. Provided written informed consent.
3. Spontaneous induced menopause as defined by one of the followings:

   * Amenorrhea of ≥12 months
   * After bilateral oophorectomy
   * FSH levels>30 IU
4. One or more VVA related symptoms (i.e., itching, dryness, burning, pain, dyspareunia, or dysuria), after other possible causes of these complaints have been excluded.
5. Characteristic atrophic changes (see above) on gynaecological examination.
6. Normal Papanicolaou (PAP) smear test from the last 3-5 years: if needed and as indicated according to the Israeli guidelines.
7. Negative urine analysis test - urine stick.
8. Asymptomatic for bacterial or fungal vaginitis.
9. Vaginal canal, introitus and vestibule free of injuries and bleeding.
10. Able and willing to comply with the treatment/ follow-up schedule and requirements.
11. Normal general gynecological exam from the last year including US.

Exclusion Criteria:

1. Vaginal Health Index Score (VHIS) < 5.
2. Active genital infection.
3. Vaginal bleeding which did not underwent evaluation.
4. Previous vulvar, vaginal or cervical dysplasia, within the last 2 years, or previous cancer.
5. Recurring urinary tract infection or recurring infection of genital herpes (≥ 3 episodes in the recent year).
6. Pelvic Organ prolapse (POP) >II, according to the pelvic organ prolapse quantification system (POP-Q).
7. Serious systemic disease or any chronic condition that could interfere with study compliance.
8. Any local, systemic and/or chronic autoimmune infection.
9. Taken part in a clinical trial concerning VVA, within 30 days prior to the enrolment.
10. Allergy to lidocaine or tetracaine.
11. Genital skin disease that may interfere with the treatment (these subjects should be included/excluded according to the investigator's discretion).
12. Use of anticoagulants, within 5 days prior to enrolment.
13. Active positive HPV test.
14. Active positive HSV (Acute or actively present within the last 2 months).
15. Heavy smoker (>1 pack of cigarettes a day)
16. Any disease or medication that may interfere with the wound healing/immune function.
17. Pregnancy / breast feeding.
18. Any other reason that, in the opinion of the investigator, prevents the subject from participating in the study or compromise the subject safety.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients that suffers from Vulvo-Vaginal Atrophy (VVA)
Enrollment: 20 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of Pixel CO2 laser (FemiLift™) for the treatment of VVA via the patient symptoms and complaints. | Two years
  The efficacy of Pixel CO2 laser (FemiLift™) treatment will be evaluate by:
  1. Improvement in VVA symptoms (itching, burning, dryness, dyspareunia, and dysuria) as evaluated by the subject, using a Numeric Rating Scales (NRSs) of 0-10.
  2. Improvement in sexual function as evaluated by the subject, using the Female Sexual Function Index (FSFI)
To evaluate gene expression following the FemiLiftTM treatment | Two years
  Changes in gene expression profile, 2 weeks following the third FemiLiftTM treatment (Tx3), compared to baseline.
  The list of genes chosen for RT PCR following a CO2 laser treatment on vaginal mucosa, includes genes taken from the following biological pathways: inflammatory response, wound healing, extracellular remodeling and connective tissue formation.

CONTACTS AND LOCATIONS:
Overall Officials: Jonia Alsheik, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel